CLINICAL TRIAL: NCT01919853
Title: Treatment for Breast and Colorectal Cancer Survivors With Persistent Cancer-Related Fatigue: A Randomized Controlled Trial
Brief Title: Treatment for Persistently Fatigued Cancer Survivors: A Randomized Controlled Trial With Biomarker Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Walther Cancer Institute (Other); Indiana Clinical and Translational Sciences Institute (Other)
Responsible Party: Principal Investigator, Shelley Johns, Assistant Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01206008951; 0106.01 (Other Grant/Funding Number: Walther Cancer Foundation, Inc.)
Record Dates: First submitted 2013-07-30; First posted 2013-08-09 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Fatigue
Keywords: Cancer; Fatigue; Mindfulness; Meditation; Neoplasms; Signs and symptoms
MeSH Terms: conditions — Fatigue; Neoplasms; Signs and Symptoms | interventions — Mindfulness-Based Stress Reduction; Educational Status; Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness-Based Stress Reduction (Experimental): The MBSR intervention is an 8-week course meeting 2 hours weekly. The curriculum is based on MBSR manuals with a brief CRF education component incorporated into the first and second class sessions, drawing from information from the National Comprehensive Cancer Network clinical practice guidelines for CRF. In general, the MBSR class includes guided meditation practice; mindful, gentle movement (hatha yoga); didactic material on self-regulatory responses to stress; and group discussion that includes the participants' growing incorporation of mindfulness in adapting to life experiences. Along with class time, each participant is asked to commit 20 minutes per day, six days per week to formal meditation practice using compact disk recordings of the teacher's voice.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Attention Control (Active Comparator): The attention control is an 8-week class meeting 2 hours weekly. The group sessions are supportive in tone, focus on pre-designated topics relevant to fatigue management (e.g., sleep hygiene, nutrition, exercise, emotional regulation), and involve weekly readings and open group discussion about session topics. This condition contains "non-specific" factors similar to MBSR (e.g., facilitator offering participants compassionate attention, empathy, genuine caring, and an opportunity to discuss what is important to them in a supportive environment); however, mindfulness is not presented/practiced in the group.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction
  Other Names: MBSR
  Arms: Mindfulness-Based Stress Reduction
Behavioral: Attention Control
  Other Names: Education/support group
  Arms: Attention Control

SUMMARY:
The purpose of this study is to compare the effects of Mindfulness-Based Stress Reduction (MBSR) to an attention control psycho-educational support group in treating cancer-related fatigue (CRF) in early-stage (0-III) post-treatment cancer survivors with clinically-significant CRF. The study will collect, store, and later analyze blood and urine samples for several biomarkers that may be linked to persistent CRF in cancer survivors.

DETAILED DESCRIPTION:
This is a randomized, attention control clinical trial to compare MBSR to support and education on biobehavioral outcomes in early-stage (0-III) post-treatment cancer survivors with clinically-significant CRF. The study will use quantitative and qualitative methods to evaluate the following:

Primary Aim 1: Determine effect size estimates of MBSR compared to attention control in reducing fatigue interference and the severity of several cancer-related symptoms immediately post-intervention and at 6-month follow-up.

Exploratory Aim 1: To identify potential moderators of intervention effects in breast cancer survivors (BCS) and colorectal cancer survivors (CRCS), such as demographic, clinical/disease characteristics, personality traits, and baseline mindfulness level.

Exploratory Aim 2: To compare levels of a number of anti- and pro-inflammatory proteins present in blood and urine between MBSR and attention control groups immediately post-intervention and 6-month follow-up, and between fatigued and non-fatigued breast cancer survivors at baseline.

ELIGIBILITY:
Inclusion Criteria for breast cancer participants:

* be age 18 or older
* live in the Indianapolis region
* have an established first-time diagnosis of non-metastatic (stages 0-III) breast cancer treated with chemotherapy and/or radiation therapy
* be in good general health (self-report)
* have clinically-significant CRF (Fatigue Symptom Inventory [FSI severity composite ≥ 4]) that has persisted for the previous 8 weeks or longer.

Inclusion Criteria for colorectal cancer participants:

* be age 18 or older
* live in the Indianapolis region
* have an established diagnosis of colorectal cancer (any stage)
* in treatment currently or previously with chemotherapy and/or radiation therapy
* have clinically-significant CRF (Fatigue Symptom Inventory [FSI severity composite ≥ 4) that has persisted for the previous 8 weeks or longer.

Exclusion Criteria for breast cancer participants:

* cancer treatment (chemotherapy, biologic response modifiers, radiation therapy, or surgery) in prior 3 months or > 5 years ago (endocrine therapy for breast cancer is allowed)
* enrollment in hospice care
* severe depression (PHQ-8 ≥ 20)
* past participation in a mindfulness meditation class and/or having an established/ongoing meditation practice

Exclusion Criteria for colorectal cancer participants:

* enrollment in hospice care
* severe depression (PHQ-8 ≥ 20)
* past participation in a mindfulness meditation class and/or having an established/ongoing meditation practice

A non-fatigued group of post-treatment BCS will also be enrolled in order to compare baseline levels of all biomarkers and all self-reported psychosocial measures between fatigued and non-fatigued BCS.

Inclusion criteria for non-fatigued BCS participants

* being age 18 or older
* having an established first-time diagnosis of non-metastatic (stage 0-III) breast cancer
* being in good general health (self-reported)
* having FSI severity composite scores of ≤ 2

Exclusion criteria for non-fatigued BCS participants

* cancer treatment (chemotherapy, biologic response modifiers, radiation therapy, or surgery) in prior 3 months or > 5 years ago (endocrine therapy for breast cancer is allowed)
* enrollment in hospice care
* severe depression (PHQ-8 ≥ 20)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in cancer-related fatigue functional interference | from baseline to 6 month follow-up
  The Fatigue Symptom Inventory interference subscale will be used to assess the degree to which CRF was judged to interfere with quality of life across seven domains over the previous week.

SECONDARY OUTCOMES:
Change in cancer-related fatigue severity | from baseline to 6 month follow-up
  The Fatigue Symptom Inventory severity subscale will be used to assess the most, least, and average fatigue in the past week, as well as current fatigue.
Change in vitality | from baseline to 6 month follow-up
  The Short Form (36) Health Survey Vitality Scale will be used to assess how much during the past 4 weeks the person had a lot of energy, felt full of life, felt worn out, and felt tired.
Change in depression | from baseline to 6 month follow-up
  The PHQ-8 scale will be used to assess how often the person has been bothered over the previous 2 weeks by symptoms of depression, including little interest or pleasure in doing things and feeling down, depressed, or hopeless.
Change in anxiety | from baseline to 6 month follow-up
  The GAD-7 scale will be used to assess how often the person has been bothered over the previous 2 weeks by symptoms such as: feeling nervous, anxious, or on edge; not being able to stop or control worrying; and trouble relaxing.
Change in sleep disturbance | from baseline to 6 month follow-up
  The Insomnia Severity Index will be used to assess the perceived severity of insomnia and the impact of sleep difficulties over the previous 2 weeks.
Change in pain | from baseline to 6 month follow-up
  The Brief Pain Inventory-3 is a brief pain measure derived from the Brief Pain Inventory. It is also known as the PEG and will be used to assess average pain intensity (P), interference with enjoyment of life (E), and interference with general activity (G) over the past week.
Change in fear of recurrence | from baseline to 6 month follow-up
  The Concerns About Recurrence Scale will be used to assess overall frequency, potential for upset, consistency, and intensity of recurrence fears.
Change in attentional function | from baseline to 6 month follow-up
  The Attentional Function Index will be used to assess perceived effectiveness in common activities requiring attention and working memory.

OTHER OUTCOMES:
Change in mindfulness | from baseline to 6 month follow-up
  The Five Facet Mindfulness Questionnaire will be used to assess the five facets of a general tendency to be mindful in daily life- observing, describing, acting with awareness, non-judgment of inner experience, and non-reactivity to inner experience.
Change in self-compassion | from baseline to 6 month follow-up
  The Self-Compassion Scale-Short Form will be used to assess attitudes associated with self-compassion. The scale includes 3 positive subscales (self-kindness, common humanity, mindfulness) and 3 negative subscales (self-judgement, isolation, and over-identification).

CONTACTS AND LOCATIONS:
Overall Officials: Shelley Johns, PsyD, Principal Investigator — Indiana University
Locations (4):
- United States (4):
  - Community Health Network--Community North and Carmel Pavilion, Carmel, Indiana
  - Indiana University, Indianapolis, Indiana
  - Invoke Yoga Studio, Indianapolis, Indiana
  - Ransburg YMCA, Indianapolis, Indiana